CLINICAL TRIAL: NCT04478773
Title: Evaluating MRI Scanning in Patients With Fractured or Abandoned Endocardial Leads
Brief Title: Adverse Events of MRI With Abandoned Leads
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to challenges with recruitment and insufficient insurance coverage for the required procedures, which prevented continuation of the trial.
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-43
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pacemaker Electrode Lead Fracture; ICD
Keywords: abandoned lead; fractured lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Patient will receive MRI
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI with or without contrast

SUMMARY:
The purpose of this study is to determine the safety and efficacy of MRI scanning in patients with fractured or abandoned endocardial leads. Specifically, the investigators aim to provide community-acquired data that can be used in Medicare and Medicaid coverage determinations and to investigate whether patients with fractured or abandoned leads can safely be scanned using an MRI and to evaluate the impact of MRI availability on patient care in this population. This study also aims to validate similar studies conducted by Mayo Clinic, the Hospital of the University of Pennsylvania and Johns Hopkins Medicine that employ MRI in the abandoned lead patient population.

ELIGIBILITY:
Inclusion criteria:

* Patients implanted with or without an ICD or pacemaker and with a fractured or an abandoned or non-functional endocardial lead, and who have a clinical need for MR imaging
* Patients are English or Spanish speaking and able to review and sign the consent

Exclusion criteria:

* Patients who complete the MRI standard screening form and are deemed inappropriate for MRI for any reason other than abandoned or fractured endocardial, or epicardial lead.
* Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events related to Magnetic Resonance Imaging (MRI) in patients with abandoned or fractured pacemaker or implantable cardioverter defibrillator (ICD) leads | 2 hours
  Incidence of symptoms and adverse events related to Magnetic Resonance Imaging (MRI) in patients with abandoned or fractured pacemaker or implantable cardioverter defibrillator (ICD) leads.
  The following measures will be collected twice during the MRI scan and reported via patient questionnaire and reported observation by technologist and electrophysiology physician or advance practice provider. Proportion/percentage of participants with:
  1. Pulling in pocket
  2. Chest pain
  3. Burning in pocket
  4. Palpitations
  5. Shortness of breath
  6. Other
  Adverse Events - collected via device monitor after MRI scan. Proportion/percentage of participants with:
  1. Atrial fibrillation
  2. Ventricular arrhythmias
  3. Frequent premature ventricular contractions with hemodynamic instability
  4. Symptomatic bradycardia with heart rate less than 40 beats per minute

SECONDARY OUTCOMES:
Understand longitudinal utilization and safety of subsequent MRIs | 7 years
  The second component of the study allows subjects to re-enroll for subsequent MRI scans as ordered by their physician to understand utilization and safety.
  The following measures will be collected and reported via patient questionnaire and reported observation by technologist and electrophysiology physician or advance practice provider :
  Patient Reported Symptoms - collected twice during the MRI scan.
  Number of participants with a subsequent MRI that experience:
  1. pulling in pocket
  2. chest pain
  3. burning in pocket
  4. palpitations
  5. shortness of breath
  6. Other
  Adverse Events - collected via device monitor after MRI scan. Number of participants with:
  1. atrial fibrillation
  2. ventricular arrhythmias
  3. frequent premature ventricular contractions with hemodynamic instability
  4. symptomatic bradycardia with heart rate less than 40 beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Bansal, MD, Principal Investigator — The Heart Group
Locations (1):
- Lancaster General Health, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04478773/Prot_000.pdf